CLINICAL TRIAL: NCT04365283
Title: Clinical Evaluation of New Bioactive Restorative Material Versus High Viscosity Glass Hybrid Reinforced Glass Ionomer in Restoration of Proximal Lesions: A Randomized Clinical Trial
Brief Title: New Bioactive Restorative Material vs GIC in Restoration of Proximal Lesions
Acronym: Bioactive
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rana Ayman Kamal (Other)
Responsible Party: Sponsor-Investigator, Rana Ayman Kamal, Resident, Conservative Dentistry Department, Faculty of Dentistry, Cairo University, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25091992
Record Dates: First submitted 2020-04-20; First posted 2020-04-28 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Randomized Clinical Trial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New Bioactive Restorative Material (Experimental): ACTIVA Presto restorative material
  Interventions: Procedure: New Bioactive Restorative Material (ACTIVA Presto)
- High Viscosity Glass Hybrid Reinforced Glass Ionomer (Active Comparator): EQUIA Forte restorative material
  Interventions: Other: High Viscosity Glass Hybrid Reinforced Glass Ionomer (EQUIA Forte)

INTERVENTIONS:
Procedure: New Bioactive Restorative Material (ACTIVA Presto) — New Bioactive Restorative Material
  Arms: New Bioactive Restorative Material
Other: High Viscosity Glass Hybrid Reinforced Glass Ionomer (EQUIA Forte) — High Viscosity Glass Hybrid Reinforced Glass Ionomer
  Arms: High Viscosity Glass Hybrid Reinforced Glass Ionomer

SUMMARY:
ACTIVA BioACTIVE products are allegedly the first dental resins with a bioactive ionic resin matrix, shock-absorbing rubberized resin component, and reactive ionomer glass fillers that mimic the physical and chemical properties of natural teeth. These bioactive materials actively participate in the cycles of ionic exchange that regulate the natural chemistry of our teeth and saliva and contribute to the maintenance of tooth structure and oral health. They are claimed to have the strength, esthetics and physical properties of composites and are more bioactive than glass ionomers, combining the best attributes of both materials without compromising either one.

DETAILED DESCRIPTION:
High caries risk patients are those who have high DMF index, high sugar intake, poor oral hygiene, inadequate salivary flow, low pH level, as well as deficient fluoride exposure.

Therefore, their management has to be adequate and proper. To overcome these setbacks, glass ionomer cements that have advantages such as similar coefficient of thermal expansion to natural tooth tissue, physicochemical adhesion to tooth structure, biocompatability, fluoride release, low shrinkage and low marginal leakage as well as anticaries properties and increased remineralization interproximally ,which is especially beneficial in high risk caries patients, have been considered as an alternative restorative material to composite and amalgam. To enhance the mechanical properties of GIs, their constituents have been modified Comparatively, resin-modified glass ionomer (RMGIs) with a longer working time, faster setting, higher early strength, and improved appearance and translucency. Unfortunately, the RMGI's mechanical properties of are different to resin composites. Progressive development of material sciences has resulted in the introduction of bioactive restorative materials. These materials can activate a tissue repair mechanism for or synthesis and elicit a response from teeth and surrounding environment. ACTIVA BioACTIVE products are allegedly the first dental resins with a bioactive ionic resin matrix, shock-absorbing rubberized resin component, and reactive ionomer glass fillers that mimic the physical and chemical properties of natural teeth. These bioactive materials actively participate in the cycles of ionic exchange that regulate the natural chemistry of our teeth and saliva and contribute to the maintenance of tooth structure and oral health. They are claimed to have the strength, esthetics and physical properties of composites and are more bioactive than glass ionomers, combining the best attributes of both materials without compromising either one.

Activa Presto light-cured material from Pulpdent is the company's latest product that features biomimicry as Activa Bioactive dual-cured material. The material diffuses fluoride, calcium, and phosphate ions that fortify the saliva and help replace essential minerals that are lost in the decay process. This highly esthetic, light-cured resin contains these ions in a stackable resin matrix that holds its shape and does not slump. This durable product is resistant to fracturing and wear, especially so on the thin areas of enamel bevels, and is indicated for all restorative procedures replacing dentin and/or enamel, anterior or posterior.

ELIGIBILITY:
Inclusion Criteria:

Proximal lesions in posterior premolars and molars and Age 20-40 years

Exclusion Criteria:

Low caries risk patients. Lack of compliance Class V in molars Systemic diseases or severe medical complications. Pregnancy. Rampant caries Disabilities

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Proximal Contact (modified USPHS criteria) | 6 months
  Ordinal(Alfa/Bravo/Charlie)
Proximal Contact (modified USPHS criteria) | 1 Year
  Ordinal(Alfa/Bravo/Charlie)

SECONDARY OUTCOMES:
Retention(modified USPHS criteria) | 6 Months
  Ordinal(Alpha/Charlie)
Retention(modified USPHS criteria) | 1 Year
  Ordinal(Alpha/Charlie)

IPD SHARING:
Plan to Share IPD: No